CLINICAL TRIAL: NCT00665288
Title: A Survey of Attitudes and Factors Associated With Successful Cardiopulmonary Resuscitation (CPR) Knowledge Transfer in an Older Population Most Likely to Witness Cardiac Arrest
Brief Title: Survey of Attitudes and Factors Associated With CPR in an Older Population
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2007751-01H
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; heart arrest; CPR; resuscitation; bystander CPR
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to conduct a survey to better understand the factors associated with undertaking cardiopulmonary resuscitation (CPR) training and performing CPR in an emergency situation.

DETAILED DESCRIPTION:
Background: Overall survival rate for out-of-hospital cardiac arrest rarely exceeds 5%. While bystander cardiopulmonary resuscitation (CPR) can increase survival for cardiac arrest victims up to four times, bystander CPR rates remain low in Canada (15%). Survivors have a quality of life similar to the general population. Most cardiac arrest victims are men in their sixties; they usually collapse in their own home (85%), where bystander CPR rates are even lower. The event is witnessed by a family member or bystander 50% of the time. These statistics appear to support a strategy of targeted CPR training for an older population that is most likely to witness a cardiac arrest event. Interest in CPR training appears to decrease with advancing age. Behaviour surrounding CPR training and performance has never been studied using the theoretical constructs of a well validated behavioural theory (the Theory of Planned Behaviour).

Objectives: The overall goal of this study is to conduct a survey to better understand the behavioural factors associated with successful CPR knowledge transfer in an independent-living older population (aged 55 or more). Specific objectives are: 1) To conduct semi-structured qualitative interviews to identify factors influencing CPR training and performance behaviours; 2) To then develop a survey instrument about factors influencing CPR training and performance behaviours based on a systematic review of the literature, the results of the semi-structured interviews, and theoretical constructs; and 3) To conduct a telephone survey among an independent-living population aged 55 or more using the survey instrument, and to identify factors and strategies that might be targeted by KT interventions.

Methods: Objective 1: We will tape-record semi-structured qualitative interviews conducted among 20 randomly selected participants aged 55 or older, and perform inductive analyses to identify categories and themes. Objective 2: The survey instrument will be developed based on a completed systematic review of the literature, and results from objective 1. The two behaviours under study will be �seeking CPR training and providing CPR to a cardiac arrest victim�. Objective 3: We will develop and conduct a nation-wide telephone survey using random digit dialling. The telephone survey will be centrally administered and stratified by province and large or small communities in order to obtain a representative random sample of the Canadian population. The study population will include all men and women aged 55 or older, living independently in the community, with the ability to communicate in English or French. We will seek to obtain a participation rate of 60% or greater. We estimate requiring approximately 500 respondents to identify factors and strategies for improving CPR KT in our target population. Analyses will include measures of sampling bias, reliability of the measures, construct validity, as well as multiple regression analyses to identify constructs and beliefs most salient to seniors� decisions about whether to attend CPR classes or perform CPR.

ELIGIBILITY:
Inclusion Criteria:

* Canadian; stratified by province
* Independent-living individuals aged 55 years or older
* Ability to communicate in French or English

Exclusion Criteria:

* persons living in the Northwest Territories, Yukon Territory, or Nunavut

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Independent-living individuals aged 55 years or older
Sampling Method: Non-Probability Sample
Enrollment: 412 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Vaillancourt C, Kasaboski A, Charette M, Islam R, Osmond M, Wells GA, Stiell IG, Brehaut JC, Grimshaw JM. Barriers and facilitators to CPR training and performing CPR in an older population most likely to witness cardiac arrest: a national survey. Resuscitation. 2013 Dec;84(12):1747-52. doi: 10.1016/j.resuscitation.2013.08.001. Epub 2013 Aug 27. PMID 23989115
- [Derived] Vaillancourt C, Charette M, Kasaboski A, Brehaut JC, Osmond M, Wells GA, Stiell IG, Grimshaw J. Barriers and facilitators to CPR knowledge transfer in an older population most likely to witness cardiac arrest: a theory-informed interview approach. Emerg Med J. 2014 Sep;31(9):700-5. doi: 10.1136/emermed-2012-202192. Epub 2013 May 1. PMID 23636603
- [Derived] Vaillancourt C, Grimshaw J, Brehaut JC, Osmond M, Charette ML, Wells GA, Stiell IG. A survey of attitudes and factors associated with successful cardiopulmonary resuscitation (CPR) knowledge transfer in an older population most likely to witness cardiac arrest: design and methodology. BMC Emerg Med. 2008 Nov 5;8:13. doi: 10.1186/1471-227X-8-13. PMID 18986547

RESULTS

PARTICIPANT FLOW:
Groups:
- CPR Training Survey: This is the group of respondents who completed the survey regarding intention to participate in CPR training.
- CPR Performing Survey: This is the group of respondents who completed the survey concerning intention to perform CPR.
Period: Overall Study
Arm/Group | CPR Training Survey | CPR Performing Survey
Started | 220 | 192
Completed | 220 | 192
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPR Training Survey | CPR Performing Survey | Total
Number analyzed (Participants) | 220 | 192 | 412
Age, Continuous [Mean (Full Range); unit: years] | 67 [55 to 88] | 66 [55 to 89] | 66 [55 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 110 | 242
  Male | 88 | 82 | 170
Region of Enrollment [Number; unit: participants]
  Canada | 220 | 192 | 412
Past CPR Training [Count of Participants; unit: Participants] | 127 | 112 | 239
Performed CPR [Count of Participants; unit: Participants] | 34 | 24 | 58

OUTCOME MEASURES:

1. Primary Outcome: Measure the Intent to Engage in CPR Training or Intent to Perform CPR
Description: Mean intention to complete CPR training in the next 6 months as well as intention to perform CPR on a victim in cardiac arrest was assessed using a 5-point Likert scale with higher scores indicating stronger intentions (1=strongly disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, 5=strongly agree).
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | CPR Training Survey | CPR Performing Survey
Number analyzed (Participants) | 220 | 192
score on a scale | 3.6 [3.4 to 3.7] | 4.1 [4.0 to 4.3]

ADVERSE EVENTS:
Arm/Group | CPR Training Survey | CPR Performing Survey
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/192
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/192
Other Adverse Events (participants affected / at risk) | 0/220 | 0/192

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No